CLINICAL TRIAL: NCT05606497
Title: OPtimal TIming of COrticosteroids in Early-onset Fetal Growth REstriction: the OPTICORE Study
Acronym: OPTICORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Stichting Achmea Gezondheidszor (Other)
Responsible Party: Principal Investigator, Dr. Judith Kooiman, Principal Investigator, UMC Utrecht
Other Study IDs: 22/613
Record Dates: First submitted 2022-10-24; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Fetal Growth Retardation
Keywords: fetal growth restriction; retrospective cohort study; antenatal corticosteroids; dynamic predictive tool
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Adrenal Cortex Hormones; Betamethasone; Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early-onset FGR
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Corticosteroid — Antenatal corticosteroids are administered to pregnancies at risk for preterm birth in order to reduce risks of neonatal morbidity and mortality following preterm birth.
  Other Names: Antenatal corticosteroids; Betamethasone; Dexamethasone

SUMMARY:
The aim of this observational study is to optimize the timing of antenatal corticosteroids administered to patients with pregnancies complicated by early-onset fetal growth restriction in order to reduce neonatal morbidity and mortality. In the Netherlands two main timing strategies of antenatal corticosteroids are commonly practiced. In this study the investigators will compare these two timing strategies regarding CCS administration in early-onset FGR on the combined endpoint of perinatal, neonatal and in-hospital mortality. In addition, the investigators aim to develop a dynamic, prediction tool, a novel technique in prediction research to predict the time-interval in days until delivery within this population. With that, the investigators aim to reduce neonatal morbidity and mortality for future FGR pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Early-onset FGR in accordance with the consensus-based definition of Gordijn et al. (19);
* Singleton pregnancy;
* Age ≥ 18 years;
* Installed active, neonatal management after counselling (thus having an indication for CCS administration in case of birth < 34 weeks of gestational age).

Exclusion Criteria:

* Multiple pregnancies;
* Fetal congenital abnormalities or antenatal diagnosed genetic disorders;
* Patients who stated that their patient or offspring data may not be used for scientific research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Singleton pregnancies complicated by early-onset FGR will be included in the study if they opt for active, neonatal management after counselling and are at least 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome for the comparison of timing strategies will be the number of perinatal, neonatal and in-hospital deaths in the offspring, assessed by scrutinizing medical records | From date of diagnosis of early-onset FGR up to hospital-discharge of the offspring, date of death of the offspring will be documented.
  This data will be validated by use of the Dutch perinatal registration data (Perined)
The primary outcome measure for the dynamic predictive tool will be defined as 'days until delivery'. | From date of diagnosis of early-onset FGR up to delivery data regarding the candidate predictors, summarized under 'Description', will be documented on every day an ultrasound examination is performed.
  Candidate predictors for the dynamic, predictive tool will be: estimated fetal weight, pulsatility index of the umbilical artery, pulsatility index of the cerebral middle artery, cerebroplacental ratio, pulsatility index of veins ductus venosus, absence of interval growth, repetitive decelerations on CTG, short-term variability, subjective fetal movements, presence of hypertensive disorders of pregnancy, use of anti-hypertensive drugs, use of magnesium sulphate, number of hypertensive crises, presence of lung edema, progression of organ dysfunction.

SECONDARY OUTCOMES:
Mode of birth, assessed by scrutinizing medical records. | This outcome measure will be documented by use of data from the day of birth.
  Mode of birth defined as vaginal or caesarian section.
Number of stillbirths, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to delivery this outcome measure will be documented.
  Stillbirth is defined as death of fetus ante- or intrapartum
Gestational age at birth (in days), assessed by scrutinizing medical records. | This outcome measure will be documented by use of data from the day of birth.
  Gestational age will be recorded in weeks as well.
Number of preterm births, assessed by scrutinizing medical records. | This outcome measure will be documented by use of data from the day of birth.
  Preterm birth defined as delivery before 37.0 weeks of gestational age.
Number of extremely preterm births, assessed by scrutinizing medical records. | This outcome measure will be documented by use of data from the day of birth.
  Extremely preterm birth is defined as delivery before 28 weeks of gestational age.
Birthweight (in grams), assessed by scrutinizing medical records. | This outcome measure will be documented by use of data from the day of birth.
  Birthweight defined as weight at time of birth (in grams)
Number of neonates with birthweight < 10th percentile (according to Hoftiezer percentiles), assessed by scrutinizing medical records. | This outcome measure will be documented by use of data from the day of birth.
Number of neonates with birthweight < 3rd percentile (according to Hoftiezer percentiles), assessed by scrutinizing medical records. | This outcome measure will be documented by use of data from the day of birth.
Number of neonates with need for mechanical ventilation, assessed by scrutinizing medical records. | From delivery up to hopsital-discharge of the offspring this outcome measure will be documented.
  Mechanical ventilation defined as need for intubation and mechanical ventilation to support gas exchange
Number of neonates diagnosed with bronchopulmonary dyspasia, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Bronchopulmonary dysplasia is diagnosed if gestational age <32 weeks: at a postmenstrual age of 36 weeks, >21% oxygen has been administered cumulatively for 28 or more days
Number of neonates diagnosed with necrotizing enterocolitis ≥ 2 according to the Bell's stages, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
Number of neonates diagnosed with neonatal seizures, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Neonatal seizures defined as transient electrographic change in the brain due to an abnormal, excessive or synchronous neuronal activity either with the occurrence of clinical signs (electro-clinical) or without them (electrographic only) in preterm infants
Number of neonates diagnosed with hypoxic-ischemic encephalopathy, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Hypoxic-ischemic encephalopathy defined as a clinical syndrome that results from a severe or prolonged hypoxic-ischemic episode before or during birth
Number of neonatal deaths, assessed by scrutinizing medical records. | From delivery up to 28 days after birth of the offspring this outcome measure will be documented.
  Death of the neonate within 28 days after birth
Number of in-hospital deaths, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Death of the neonate until hospital-discharge
Number of neonates diagnosed with respiratory distress syndrome, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Neonatal respiratory distress syndrome, characterized by extensive lung inflammation and surfactant catabolism leading to lung dysfunction, with need for surfactant
Number of neonates diagnosed with intraventricular hemorrhage, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Intraventricular hemorrhage grade 3 according to Papile et al., venous infarction, posthemorrhagic ventricular dilatation needing treatment
Number of neonates diagnosed with cystic periventricular leukomalacia, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Cystic periventricular leukomalacia is characterized by diffuse injury of the white matter, which possibly leads to cerebral palsy
Number of neonates diagnosed with retinopathy of prematurity, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Retinopathy of prematurity with plus disease for which treatment is needed
Number of neonates diagnosed with neonatal sepsis, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Distinction will be made in early-onset vs late-onset and clinical vs culture-proven
Number of neonates diagnosed with persistent pulmonary hypertension of the newborn, assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
  Persistent pulmonary hypertension of the newborn occurs in case of persistent abnormally, elevated pulmonary vascular resistance after birth, leading to severe hypoxemia
Duration of supplemental oxygen therapy during admission of the offspring (in days), assessed by scrutinizing medical records. | From delivery up to hospital-discharge of the offspring this outcome measure will be documented.
Number of neonates with need for mechanical ventilation < 72 hours post-partum, assessed by scrutinizing medical records. | From delivery up to 72 hours after birth this outcome measure will be documented.
  This is defined as need for intubation and mechanical strategies to support gas exchange within 72 hours after birth
Number of childs with cognitive impairment, assessed by scrutinizing medical records. | From delivery up to 24 months corrected age of the offspring this outcome measure will be documented.
  A decreased ability of cognitive function using Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) at a corrected age of 24 months,. Severe disability will be defined as a Bayley Mental Development Index score more than 2SD below the mean score (i.e. ≤70). Moderate disability will be defined as a Bayley Mental Development Index score 1 to 2 SD below the mean score (i.e. 71-85)
Number of childs with motor impairment, assessed by scrutinizing medical records. | From delivery up to 24 months corrected age of the offspring this outcome measure will be documented.
  A decreased ability of fine and gross motor function using part of the Bayley Scales and Infant and Toddler Development, Third Edition (BSID-III) at corrected age of 24 months. Severe disability will be defined as a score of more than 2 SD below the mean score (i.e. ≤70). Moderate disability will be defined as a score 1 to 2SD below the mean score (i.e. 71-85)
Number of childs diagnosed with cerebral palsy, assessed by scrutinizing medical records. | From delivery up to 24 months corrected age of the offspring this outcome measure will be documented.
  Cerebral palsy is a group of disorders of the development of movement and posture, causing activity limitation, that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain
Number of childs with hearing impairment, assessed by scrutinizing medical records. | From delivery up to 24 months corrected age of the offspring this outcome measure will be documented.
  A decreased ability of the auditory system requiring hearing aids or deafness
Number of childs with visual impairment, assessed by scrutinizing medical records. | From delivery up to 24 months corrected age of the offspring this outcome measure will be documented.
  A decreased ability of the visual system requiring aids or blindness
Number of maternal deaths, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of patients diagnosed with (pre-)eclampsia, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with a Glasgow Coma Score < 13, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with a stroke or reversible ischaemic neurological deficit, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with a transient ischaemic attack, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with cortical blindness or retinal detachment, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with posterior reversible encephalopathy, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with need for positive inotropic support, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with need for infusion of a third parenteral antihypertensive drug, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with myocardial ischaemia or infarction, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with oxygen saturation below 90%, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with ≥ 50% fraction of inspired oxygen for more than one hour, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with need for intubation, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with pulmonary oedema, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
  Determined by pulmonary auscultation.
Number of mothers with need for transfusion of any blood product, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with a platelet count < 50x10^9 per liter with no transfusion, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with hepatic dysfunction, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
  Hepatic dysfunction defined as asparate aminotransferase and alanine aminotransferase elevated more than twice the upper limit of normal.
Number of mothers with hepatic haematoma or rupture, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers with acute renal insufficiency, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
  Acute renal insufficiency defined as creatinine >150 μmol/L with no pre-existing renal disease.
Number of mothers with acute renal failure, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
  Acute renal failure defined as creatinine >200 μmol/L in patients with pre-existing renal disease.
Number of mothers with need for renal dialysis, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with placental abruption, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with severe ascites, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.
Number of mothers diagnosed with Bell's palsy, assessed by scrutinizing medical records. | From diagnosis of early-onset FGR up to six weeks post-partum this outcome measure will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: J. Kooiman, MD, PhD, Epidemiologist, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Wilhelmina Children's Hospital, Utrecht, Netherlands

REFERENCES:
- [Derived] van de Meent M, Kleuskens DG, Ganzevoort W, Gordijn SJ, Kooi EMW, Onland W, van Rijn BB, Duvekot JJ, Kornelisse RF, Al-Nasiry S, Jellema RK, Knol HM, Manten GTR, Mulder-de Tollenaer SM, Derks JB, Groenendaal F, Bekker MN, Schuit E, Lely AT, Kooiman J. OPtimal TIming of antenatal COrticosteroid administration in pregnancies complicated by early-onset fetal growth REstriction (OPTICORE): study protocol of a multicentre, retrospective cohort study. BMJ Open. 2023 Mar 17;13(3):e070729. doi: 10.1136/bmjopen-2022-070729. PMID 36931680